CLINICAL TRIAL: NCT03520647
Title: Haplo-identical Transplantation for Severe Aplastic Anemia, Hypo-plastic MDS and PNH Using Peripheral Blood Stem Cells and Post-transplant Cyclophosphamide for GVHD Prophylaxis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180090; 18-H-0090
Record Dates: First submitted 2018-05-09; First posted 2018-05-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Severe Aplastic Anemia (SAA); Hypo-Plastic Myelodysplastic Syndrome (MDS); Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: Haploidentical CD34+cells; Non-Myeloablative
MeSH Terms: conditions — Anemia, Aplastic; Hemoglobinuria, Paroxysmal | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): G-CSF mobilized peripheral stem cells and post haplo-identical transplantation cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Other: Peripheral Blood Stem Cells

INTERVENTIONS:
Drug: Cyclophosphamide — This research protocol is therefore designed to evaluate the safety and effectiveness of using an unmanipulated G-CSF mobilized peripheral stem cell allograft from a haploidentical donor and post-transplant cyclophosphamide for patients with SAA, or SAA evolving to MDS, or PNH that has proven to be refractory to conventional immunosuppressive therapy (IST) in patients who lack an HLA-matched donor (sibling/ or matched unrelated donor.
Other: Peripheral Blood Stem Cells — This research protocol is therefore designed to evaluate the safety and effectiveness of using an unmanipulated G-CSF mobilized peripheral stem cell allograft from a haploidentical donor and post-transplant cyclophosphamide for patients with SAA, or SAA evolving to MDS, or PNH that has proven to be refractory to conventional immunosuppressive therapy (IST) in patients who lack an HLA-matched donor (sibling/ or matched unrelated donor.

SUMMARY:
Background:

Severe aplastic anemia (SAA), and myelodysplastic syndrome (MDS), and paroxysmal nocturnal hemoglobinuria

(PNH) cause serious blood problems. Stem cell transplants using bone marrow or blood plus chemotherapy can help. Researchers want to see if using peripheral blood stem cells (PBSCs) rather than bone marrow cells works too. PBSCs are easier to collect and have more cells that help transplants.

Objectives:

To see how safely and effectively SAA, MDS and PNH are treated using peripheral blood hematopoietic stem cells from a family member plus chemotherapy.

Eligibility:

Recipients ages 4-60 with SAA, MDS or PNH and their relative donors ages 4-75

Design:

Recipients will have:

* Blood, urine, heart, and lung tests
* Scans
* Bone marrow sample

Recipients will need a caregiver for several months. They may make fertility plans and a power of attorney.

Donors will have blood and tissue tests, then injections to boost stem cells for 5-7 days.

Donors will have blood collected from a tube in an arm or leg vein. A machine will separate stem cells and maybe white blood cells. The rest of the blood will be returned into the other arm or leg.

In the hospital for about 1 month, recipients will have:

* Central line inserted in the neck or chest
* Medicines for side effects
* Chemotherapy over 8 days and radiation 1 time
* Stem cell transplant over 4 hours

Up to 6 months after transplant, recipients will stay near NIH for weekly physical exams and blood tests.

At day 180, recipients will go home. They will have tests at their doctor s office and NIH several times over 5 years.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA),myelodysplastic syndrome (MDS), and paroxysmal nocturnal hemoglobinuria (PNH) are life-threatening bone marrow disorders. For SAA patients, long term survival can be achieved with immunosuppressive treatment. However, of those patients treated with immunosuppressive therapy, one quarter to one third will not respond, and about 50% of responders will relapse.

Although allogeneic stem cell transplantation (allo-SCT) offers the opportunity of cure, HLA-matched donors are available for only half the patients needing a transplant. Combined haplo-cord transplantation has recently been shown to be a viable transplant option for those patients lacking an HLA matched donor. In our ongoing protocol 08-H-0046, we have utilized this approach in 29 patients with SAA, and SAA evolving to MDS with 27/29 patients having sustained engraftment and achieving transfusion independence. However, engraftment patterns have varied substantially and, in some patients,, cord engraftment was profoundly delayed or never occurred.

Haploidentical peripheral blood stem cell transplantation (haplo-SCT) has the advantage over cord transplantation of immediate allograft availability, higher stem cell doses, and the feasibility of repeating cell collections if necessary for collecting CD34+ cells for stem cells boosts or lymphocytes to treat or prevent disease relapse or infection. Recently, the use of post-transplant cyclophosphamide (Cy) has been shown to be an effective strategy to prevent GVHD in recipients of haploidentical HSCT, but most reports have focused on patients with hematological malignancies. At present, few data exist on the use of haploidentical transplantation using post-transplant cyclophosphamide for patients with aplastic anemia that have ATG-refractory disease and are heavily-transfused and HLA-alloimmunized. These patients are at an exceedingly high-risk for graft rejection compared to other patient populations.

This research protocol is therefore designed to evaluate the safety and effectiveness of using an unmanipulated GCSF mobilized peripheral stem cell allograft from a haploidentical donor and post-transplant cyclophosphamide for patients with SAA,SAA evolving to MDS, or PNH that has proven to be refractory to conventional therapy in patients who lack an HLA-matched donor (sibling/ or matched unrelated donor).

The primary endpoint of the study is chronic GVHD-free survival (defined as the percentage of patients who are alive with no evidence of moderate or severe chronic GVHD at 1-year post-transplant). Secondary endpoints will include engraftment, 100 day and 200-day treatment related mortality (TRM), and standard transplant outcome variables such as non-hematologic toxicity, incidence and severity of acute and chronic GVHD, and relapse of disease. Health related quality of life will also be assessed as secondary outcome measure.

ELIGIBILITY:
* INCLUSION CRITERIA - RECIPIENT:
* Diagnosed with severe aplastic anemia with bone marrow cellularity <30% (excluding lymphocytes) associated with RBC or platelet transfusion dependence and/or neutropenia (absolute neutrophil count less than or equal to 1000 cells/ microL or for patients receiving granulocyte transfusions, absolute neutrophil count less than or equal to 1000 cells/microL before beginning granulocyte transfusions).

OR

--History of severe aplastic anemia transformed to MDS. that meet the following criteria: a) International Prognostic Scoring System (IPSS) risk category of INT-1 or greater, b) <5% myeloblasts and <30% of cellularity in the bone marrow on screening morphologic analysis.

OR

* PNH that is either refractory to treatment with eculizumab/ravulizumab or occurs in patients who don t have access to treatment with eculizumab associated with either a) life- threatening thrombosis and/or b) cytopenia associated with transfusion dependence and/or c) recurrent and debilitating hemolytic crisis.

  * Subjects with severe aplastic anemia, hypoplastic MDS or PNH with associated bone marrow failure syndromes who have intolerance of or failure to respond to standard immunosuppressive therapy.
  * Availability of at least one HLA- haploidentical related donor (i.e. >= 5/10 HLA match: HLA-A, B, C, DR, and DQ loci) to serve as a stem cell donor for the allogeneic transplant.
  * Availability of a backup stem cell source in the event of graft rejection:
* at least one additional haploidentical related alternative donor (i.e. HLA- haploidentical related donor (i.e. >= 5/10 HLA match: HLA-A, B, C, DR, and DQ loci) or >= 9/10 HLA matched unrelated donor who is available to serve as a stem cell donor for a salvage allogeneic transplant in the event that the haplotransplant has been rejected.
* umbilical cord blood unit/s that can be used for a salvage cord blood transplant in the event that the haplo-transplant has been rejected

  * The patient does not have any HLA antibodies detectable against any of the mismatched HLA alleles expressed by the haplo-donor.
  * Ages 4-60 years inclusive.
  * Ability to comprehend the investigational nature of the study and provide informed consent. The procedure will be explained to subjects aged 4-17 years with formal consent being obtained from parents or legal guardian.

EXCLUSION CRITERIA - RECIPIENT (ANY OF THE FOLLOWING):

* Availability of an HLA identical (12/12) matched related or unrelated donor who is available within optimal timeline and suitable considering graft source and established donor selection factors (e.g. age, sex, viral exposure, ABO compatibility, pregnancy status, etc) per PI discretion.
* The patient is deemed to be a candidate for a 12/12 HLA matched unrelated stem cell transplant (availability of a donor and resources required for such a transplant).
* ECOG performance status of 2 or more.
* Major anticipated illness or organ failure incompatible with survival from transplant.
* Current pregnancy, or unwillingness to take oral contraceptives or use a barrier method of birth control or practice abstinence to refrain from pregnancy, if of childbearing potential for one year.
* HIV positive.
* Diagnosis of Fanconi s anemia (by chromosome breakage study).
* Diffusion capacity of carbon monoxide (DLCO) <40% using DLCO corrected for Hgb or lung volumes (patients under the age of 10 may be excluded from this criterion if they have difficulty performing the test correctly and thus are unable to have their DLCO assessed).
* Left ventricular ejection fraction <40% (evaluated by ECHO)
* Transaminases > 5x upper limit of normal.
* Direct bilirubin >3 mg/dl.
* Creatinine clearance < 50 cc/min/BSAm2 by 24-hour urine collection adjusted by body surface area.
* Serum creatinine > 2.5 mg/dl
* Presence of an active infection not adequately responding to appropriate therapy.
* History of a malignant disease liable to relapse or progress within 5 years.

INCLUSION CRITERIA - DONOR:

Donor deemed suitable and eligible, and willing to donate, per clinical evaluations who are additionally willing to donate blood for research. Donors will be evaluated in accordance with existing Standard NIH Policies and Procedures for determination of eligibility and suitability for clinical donation. Note that participation in this study is offered to all donors, but is not required for a donor to make a stem cell donation, so it is possible that not all donors will enroll onto this study.

EXCLUSION CRITERIA - RELATED DONOR:

None

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate 1 year chronic GVHD-free survival rate | one-year
  evaluate 1 year chronic GVHD-free survival rate (defined by the percentage of patients who are alive with no evidence of moderate or severe chronic GVHD at 1 year) of using G-CSF mobilized peripheral stem cells and post haplo-identical transplantation cyclophosphamide in subjects with severe aplastic anemia or refractory anemia (RA) or SAA subjects

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0090.html